CLINICAL TRIAL: NCT02056418
Title: A Randomized, Controlled, Single-blind Study of Effects of Enteral Nutrition and Corticosteroid on Intestinal Flora in Induction Remission of Crohn Disease in Adult
Brief Title: Effects of Enteral Nutrition and Corticosteroid on Intestinal Flora in Induction Remission of Crohn Disease in Adult
Acronym: EN
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Jinling Hospital, China (Other)
Responsible Party: Principal Investigator, Zhu Weiming, professor, Jinling Hospital, China
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ECDB-1
Record Dates: First submitted 2014-01-24; First posted 2014-02-06 (Estimated); Last update posted 2014-02-06 (Estimated); Status verified 2014-02

CONDITIONS: Crohn Disease
MeSH Terms: conditions — Crohn Disease | interventions — Enteral Nutrition; Adrenal Cortex Hormones; Prednisone; Hydrocortisone

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- enteral nutrition (Experimental): The patients receive treatment of enteral nutrition only.
  Interventions: Dietary Supplement: enteral nutrition
- Corticosteroid (Experimental): The patients receive treatment of corticosteroid only.
  Interventions: Drug: corticosteroid
- Healthy control (No Intervention): healthy people applied with normal diet.

INTERVENTIONS:
Dietary Supplement: enteral nutrition — enteral nutrition only (Nutrison Fibre, 20-30kcal/kg/day)
  Arms: enteral nutrition
Drug: corticosteroid — corticosteroid(equal dose to prednisone 0.75mg/kg/day,4 weeks)
  Other Names: prednisone; hydrocortisone
  Arms: Corticosteroid

SUMMARY:
The pathogenesis of Crohn Disease (CD) is unknown, but there is evidence show that the inadequate immune response or overreaction of the immune system against food antigens or components of the commensal flora involve it. Corticosteroid therapy is effective for adult patients with CD, but it has side effects and can't promote mucosal healing. In recent years, Enteral nutrition (EN) is becoming primary therapy in induction and maintenance remission of CD, especially in children. But the mechanism of EN in induction and maintenance remission of CD is still unclear, and parts of patient have good clinical response to EN therapy while other don't. So we design the study to explore whether EN treats CD by effecting intestinal flora and whether the intestinal flora of patient with CD relates with clinical response.

DETAILED DESCRIPTION:
The pathogenesis of CD is unknown, but there is evidence show that the inadequate immune response or overreaction of the immune system against food antigens or components of the commensal flora involve it. Corticosteroid therapy is effective for adult patients with CD, but it has side effects and can't promote mucosal healing. In recent years, EN is becoming primary therapy in induction and maintenance remission of CD, especially in children. But the mechanism of EN in induction and maintenance remission of CD is still unclear, and parts of patient have good clinical response to EN therapy while other don't. So we design the study to explore whether EN treats CD by effecting intestinal flora and whether the intestinal flora of patient with CD relates with clinical response.

ELIGIBILITY:
Inclusion Criteria:

1. Patients should be in the age range of 18 - 75 years;
2. Patients should have clinical, imaging, endoscopic and histological diagnosis of CD based on WHO criteria
3. Patients should have a CDAI score of more than 150 and have a CRP level of more than 10mg/L at enrollment;
4. Patients will not be excluded if they have received 5-ASA(Aminosalicylic acid) or immunomodulator for >8 weeks and the dose is stable
5. Informed consent

Exclusion Criteria:

1. Patients who can't tolerate enteral nutrition because of complications, such as complete intestinal obstruction, gastrointestinal perforation or bleeding etc.
2. Patients who receive corticosteroids or enteral nutrition or prebiotics /probiotics/synbiotics/antibiotic treatment in the previous 4 weeks.
3. Patients who accompanied extra-intestinal manifestations, serve complications, and active perianal disease and need other drug therapies.
4. Patients who had ostomy or colectomy or subtotal colectomy
5. Patients with end-stage disease or is expected likely to die during the study
6. Patients are participating in other clinical trials or participated within 6 months prior to this study

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2014-01; Primary Completion 2016-01 (Estimated); Study Completion 2016-01 (Estimated)

PRIMARY OUTCOMES:
change of intestinal flora of stool | 6 weeks
  Change from baseline in diversity and composition of intestinal flora of stool every week and time point of clinical remission after intervention

SECONDARY OUTCOMES:
biochemical indexes | 6 weeks
  Change from baseline of hematological and biochemical indexes (CRP(C-reactive protein), PCT(procalcitonin), ESR(erythrocyte sedimentation rate), Alb) of blood every week
CDAI(Crohn's disease activity index) | 6 weeks
  Change from baseline of CDAI every week
Fecal Calcium Protein | 6 weeks
  Change from Baseline in Fecal Calcium Protein in every week

CONTACTS AND LOCATIONS:
Locations (1):
- Department of General Surgery, Jinling hosptal,Medical School of Nanjing University, Nanjing, Jiangsu, China

REFERENCES:
- [Derived] Guo D, Fang L, Liu R, Li Y, Lv L, Niu Z, Chen D, Zhou Y, Zhu W. Exploring Different Effects of Exclusive Enteral Nutrition (EEN) and Corticosteroids on the Gut Microbiome in Crohn's Disease Based on a Three-Stage Strategy. Gastroenterol Res Pract. 2022 Jul 27;2022:6147124. doi: 10.1155/2022/6147124. eCollection 2022. PMID 35935714